CLINICAL TRIAL: NCT04570176
Title: Clinical Trial Protocol of Primary Study on Efficacy and Safety of Telesurgery for Patients With Tumors of the Urinary System Using Chinese Independently Developed "MicroHand" Surgical Robot System
Brief Title: Efficacy and Safety of Clinical Telesurgery Using Chinese Independently Developed Surgical Robot System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Haitao Niu, MD, Professor Haitao Niu, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDWG-NST600S-YCSS
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2020-09

CONDITIONS: Renal Cell Carcinoma; Bladder Cancer; Adrenal Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Adrenal Gland Neoplasms | interventions — Adrenalectomy; Cystectomy; Nephrectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urologic tumor group (Experimental): patients with adrenal adenoma, muscle-invasive bladder cancer or renal cell carcinoma are included in the experiment.
  Interventions: Procedure: adrenalectomy for adrenal adenoma

INTERVENTIONS:
Procedure: adrenalectomy for adrenal adenoma — adrenalectomy， cystectomy and nephrectomy
  Other Names: cystectomy for muscle-invasive bladder cancer; nephrectomy for patients with renal cell carcinoma.

SUMMARY:
One-arm clinical trial was adopted in this study. The surgeons performed remote urological surgery for patients through domestically produced "MicroHand" surgical robot system (Shandong Weigao Co., Ltd). The "MicroHand" surgical robot system consists of two physically separated subsystems named the "surgeon console" and "patient side cart". The surgeon console includes a stereo image viewer, two master manipulators, a control panel and several foot pedals. The patient side cart includes a passive arm that can slide in the up-down direction and be adjusted forward and backward, a swivel head that can rotate around the vertical axis, and three slave arms (one for the endoscopic camera and the other two for surgical instruments). The surgeon console (based in Qingdao) takes the surgeon's input and translates it into a control signal. After network transmission, the patient side cart (based in Anshun) translates the control signal into actual instrument manipulation. The 3D images captured by the endoscopic camera were simultaneously sent back to the screen of the surgeon console as visual feedback. Data between the surgeon console and the patient side cart were transmitted through a 5G network. The safety and effectiveness of the robotic system in remote clinical diagnosis and treatment were verified by the main judgment criterion and secondary judgment criterion. Six patients are planned to enroll in the clinical trial.

Main judgment criterion:

The robot-assisted telesurgery did not transfer to other types of surgery, such as open surgery or normal robot-assisted surgery.

Secondary judgment criterion:

operative time, blood loss, postoperative pain, preoperative adjusting time and hospitalization time.

Patient enrollment:

This trial aims to explore the safety and effectiveness of the domestically produced robotic system in remote clinical diagnosis and treatment through 5G network. Six patients are planned to enroll in the clinical trial, including 2 patients with adrenal tumor, 2 patients with bladder cancer and 2 patients with renal cell carcinoma.

DETAILED DESCRIPTION:
Objective： This clinical trial aims to evaluate the efficacy and safety of telesurgery for patients with tumors of the urinary system using Chinese independently developed "MicroHand" Surgical Robot System through 5G network.

Content： One-arm clinical trial was adopted in this study. The product was domestically produced "MicroHand" surgical robot system (Shandong Weigao Co., Ltd). Before entering the clinical study, the patients were fully informed and the written informed consent were signed. According to the inclusion criteria and exclusion criteria, the researchers will conduct a detailed screening to determine whether they are suitable for the clinical study. Telesurgery would be conducted for patients who met the inclusion criteria using "MicroHand" surgical robot system. Data between the surgeon console and the patient side cart were transmitted through a 5G network. The safety and efficacy of the robotic system in remote clinical diagnosis and treatment were verified according to the main judgment criterion and secondary judgment criterion.

Background： With the combination of robotic and network communication technology, telesurgery has become a reality. On the one hand, telesurgery can conserve and optimize medical resources, providing high-quality medical services to unbalanced areas, such as rural areas, stricken areas and battlefields. On the other hand, telesurgery can reduce the time spent by patients waiting for treatment and thus prevent diseases from worsening.

The unbalanced distribution of medical resources has been a prominent problem in China. In addition, the vast territory and relatively lower medical distribution ratio per capita make it difficult for patients to receive timely and high-quality treatment, especially those in remote and underdeveloped areas. Therefore, telesurgery is more significant in China. In recent years, surgical robot systems and network communication technology have experienced breakthroughs. The operation systems of the Da Vinci robot in America, the REVO-I robot in South Korea and the ALF-X robot in Italy are more flexible and intelligent, performing well in surgical procedures. The "Micro Hand S" system robot, independently developed in China, represents a new generation of surgical robot systems. In addition to the flexible and intelligent characteristics of traditional robots, it has a series of advantages, such as a clear interface, light weight, low cost in terms of use and maintenance, and strong equipment compatibility. After preliminary experiments, it has been successfully applied in clinical surgery6. Meanwhile, in the field of network communication, the emerging 5G mobile communication technology (the 5th generation of wireless systems, 5G technology for short) is the latest generation of cellular mobile communication technology. It is also an extension of 4G (LTE-A or WiMax), 3G (UMTS or LTE) and 2G (GSM) technology. 5G technology has a high data rate, low latency, high throughput, equipment connection on a large scale, low cost and low energy consumption. The emergence of 5G technology offers more opportunities for the prevalence of telesurgery.

In September 2019, our research group carried out the first 5G remote telesurgery using the "Micro Hand S" system robot and a 5G network between Qingdao, Shandong Province, and Xixiu, Guizhou Province, in September 2019 in China (the network communication distance was nearly 3000 km). Specifically, the investigators conducted four ultra-remote laparoscopic surgeries, including left nephrectomy, partial hepatectomy, cholecystectomy and cystectomy in a swine model under the 5G network using a domestically produced "Micro Hand S" surgical robot. the investigators accomplished four laparoscopic telesurgeries successfully, with an average network delay of 264 ms (including a round-trip transporting delay of 114 ms and a 1.20% data package loss ratio). Moreover, the total blood loss was 25 ml and no complications occurred during the procedures. The investigators demonstrated that ultra-remote laparoscopic telesurgery can be performed safely and smoothly under the 5G network using domestically produced equipment. On such basis, our research group planned to carry out this clinical trial to evaluate the efficacy and safety of telesurgery for patients with tumors of the urinary system using Chinese independently developed "MicroHand" Surgical Robot System through 5G network.

Introduction of the "MicroHand" surgical robot： The "MicroHand" surgical robot system consists of two physically separated subsystems named the "surgeon console" and "patient side cart". The surgeon console includes a stereo image viewer, two master manipulators, a control panel and several foot pedals. The patient side cart includes a passive arm that can slide in the up-down direction and be adjusted forward and backward, a swivel head that can rotate around the vertical axis, and three slave arms (one for the endoscopic camera and the other two for surgical instruments). The surgeon console (based in Qingdao) takes the surgeon's input and translates it into a control signal. After network transmission, the patient side cart (based in Anshun) translates the control signal into actual instrument manipulation. The 3D images captured by the endoscopic camera were simultaneously sent back to the screen of the surgeon console as visual feedback.

Steps of the procedure：

① The surgeon console was placed in Qingdao, Shangdong Province, while the patient side cart was placed in Anshun, Guizhou Province.

② Connections between the surgeon console and the patient side cart were established through a public 5G wireless network. Special 5G customer premise equipment (CPE) was used as a signal repeater station and amplifier. Upload and download speed will be tested as network bandwidth.

③ After general anesthesia, the supine position was maintained, the surgical area was disinfected, and pneumoperitoneum was established from the left side of the umbilicus by using a Veress needle. Then, trocars were inserted, and slave arms were delivered. Slave arm A was equipped with robotic grasp pliers, and Slave arm C was equipped with an ultrasonic scalpel (bipolar pliers or electrocautery). Robot-assisted telesurgeries, including adrenalectomy, cystectomy and nephrectomy, were performed by surgeons from the departments of urology. Surgeons in Qingdao performed the dissection and coagulation of the target organs, while assistants in Anshun performed exposure of structures and clip application. Trocar placement and position of the patients were also adjusted in each telesurgery by the assistants if necessary. After completion of the dissection, the target organs were removed by the assistant bedside. Then the pneumoperitoneum was exsufflated and the incisions were closed. Intraoperative network latencies and vital signs were monitored constantly. The master-slave manipulation consistency was assessed subjectively. The operative time, blood loss and complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-III
* BMI: 18-30Kg/m2
* adrenal tumors that need adrenalectomy (hormonally active or grow more than 1cm during annual evaluation； other benign adrenal tumors)
* patients with Robson Stage I or II renal cell carcinoma that need radical nephrectomy
* patients with Clinical Stage I or II bladder cancer that need radical cystectomy

Exclusion Criteria:

* women during pregnancy or lactation period
* patients with uncontrolled hypertension
* patients with a history of epilepsy or psychosis
* patients with severe cardiovascular disease (NYHA, grade III-IV)
* patients with cerebrovascular disease (CVD)
* patients with other diseases that cannot tolerate surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
success rate of the telesurgery | during the procedure
  The success of the telesurgery is the robot-assisted telesurgery did not transfer to other types of surgery， such as open surgery or normal robot-assisted surgery. The number of the success divided by the total number is the success rate.

SECONDARY OUTCOMES:
operative time | during the procedure
  duration of each surgery
blood loss | during the procedure
  blood loss of each surgery
latency time | during the procedure
  Mechanical response delay of the robot, endoscope imaging and image processing delay plus video codec delay equals the total delay.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Niu, PhD, Study Chair — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nguan C, Miller B, Patel R, Luke PP, Schlachta CM. Pre-clinical remote telesurgery trial of a da Vinci telesurgery prototype. Int J Med Robot. 2008 Dec;4(4):304-9. doi: 10.1002/rcs.210. PMID 18803341
- [Result] Sterbis JR, Hanly EJ, Herman BC, Marohn MR, Broderick TJ, Shih SP, Harnett B, Doarn C, Schenkman NS. Transcontinental telesurgical nephrectomy using the da Vinci robot in a porcine model. Urology. 2008 May;71(5):971-3. doi: 10.1016/j.urology.2007.11.027. Epub 2008 Mar 4. PMID 18295861
- [Result] Clayman RV. Transatlantic robot-assisted telesurgery. J Urol. 2002 Aug;168(2):873-4. No abstract available. PMID 12136861
- [Result] Marescaux J, Leroy J, Rubino F, Smith M, Vix M, Simone M, Mutter D. Transcontinental robot-assisted remote telesurgery: feasibility and potential applications. Ann Surg. 2002 Apr;235(4):487-92. doi: 10.1097/00000658-200204000-00005. PMID 11923603
- [Result] Garcia P, Rosen J, Kapoor C, Noakes M, Elbert G, Treat M, Ganous T, Hanson M, Manak J, Hasser C, Rohler D, Satava R. Trauma Pod: a semi-automated telerobotic surgical system. Int J Med Robot. 2009 Jun;5(2):136-46. doi: 10.1002/rcs.238. PMID 19222048
- [Result] Lefranc M, Peltier J. Evaluation of the ROSA Spine robot for minimally invasive surgical procedures. Expert Rev Med Devices. 2016 Oct;13(10):899-906. doi: 10.1080/17434440.2016.1236680. Epub 2016 Sep 30. PMID 27649314
- [Result] Abdel Raheem A, Troya IS, Kim DK, Kim SH, Won PD, Joon PS, Hyun GS, Rha KH. Robot-assisted Fallopian tube transection and anastomosis using the new REVO-I robotic surgical system: feasibility in a chronic porcine model. BJU Int. 2016 Oct;118(4):604-9. doi: 10.1111/bju.13517. Epub 2016 May 26. PMID 27123543
- [Result] Fanfani F, Monterossi G, Fagotti A, Rossitto C, Gueli Alletti S, Costantini B, Gallotta V, Selvaggi L, Restaino S, Scambia G. The new robotic TELELAP ALF-X in gynecological surgery: single-center experience. Surg Endosc. 2016 Jan;30(1):215-21. doi: 10.1007/s00464-015-4187-9. Epub 2015 Apr 4. PMID 25840895
- [Result] Moglia A, Ferrari V, Morelli L, Ferrari M, Mosca F, Cuschieri A. A Systematic Review of Virtual Reality Simulators for Robot-assisted Surgery. Eur Urol. 2016 Jun;69(6):1065-80. doi: 10.1016/j.eururo.2015.09.021. Epub 2015 Oct 1. PMID 26433570
- [Result] Yi B, Wang G, Li J, Jiang J, Son Z, Su H, Zhu S, Wang S. Domestically produced Chinese minimally invasive surgical robot system "Micro Hand S" is applied to clinical surgery preliminarily in China. Surg Endosc. 2017 Jan;31(1):487-493. doi: 10.1007/s00464-016-4945-3. Epub 2016 May 18. PMID 27194259
- [Result] Yi B, Wang G, Li J, Jiang J, Son Z, Su H, Zhu S. The first clinical use of domestically produced Chinese minimally invasive surgical robot system "Micro Hand S". Surg Endosc. 2016 Jun;30(6):2649-55. doi: 10.1007/s00464-015-4506-1. Epub 2015 Aug 21. PMID 26293795